CLINICAL TRIAL: NCT01999790
Title: Comparison Study Between Two Techniques for Correction of Upper Lid Retraction in Patients With Grave's Orbitopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Allan Christian Pieroni Goncalves, staff, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: protocoloretracao
Record Dates: First submitted 2013-11-17; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Graves Ophthalmopathy
Keywords: upper lid; exophthalmos; grave's orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy; Exophthalmos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blepharothomy (Experimental): Patients treated with blepharotomy to correct upper lid retraction secondary to Grave's orbitopathy
  Interventions: Procedure: blepharotomy
- posterior approach (Experimental): Patients treated with a posterior approach to correct upper lid retraction secondary to Grave's orbitopathy
  Interventions: Procedure: posterior approach

INTERVENTIONS:
Procedure: blepharotomy — upper eyelid surgery by blepharotomy
  Arms: Blepharothomy
Procedure: posterior approach — upper eyelid surgery by posterior approach
  Arms: posterior approach

SUMMARY:
Grave's ophthalmopathy is the most common cause of orbital disease in adults. The clinical presentation may vary between sub clinic symptoms to severe ones. The eyelid retraction is one of the most important signs of Grave's ophthalmopathy and can lead to cosmetic and functional problems.

The eyelid retraction can be found in the inflammatory stage and in the chronic disease, when it is stable. It can be described when the upper lid is contouring the superior limbus or positioned above that. This condition can lead to dry eye symptoms, exposure keratitis and cosmetic issues. The treatment can may be surgical or medical.

The medical treatment are usually based on controlling thyroid function and in the use of steroids, both are not specific for the lid retraction, but for the inflammation that is common in the disease.

In the longstanding disease, surgery is the most efficient treatment. There are several described techniques, they are based on the concept of weakening the muscles that act on lid elevation (levator and Muller Muscle).

Basically the techniques can be divided in two groups: the first with an anterior approach (with skin scar in the lid sulcus) and the second using a posterior approach (through the conjunctiva).

In the literature there is no consensus in deciding the best technique, regarding cosmetic results, incidence of complications, hypo or hypercorrection.

In this trial we propose to compare two distinct techniques that are already in clinical use. The blepharotomy uses a cutaneous approach and the other a conjunctival approach.

The patients will be divided in two randomized groups and surgical expected outcomes, cosmetics outcomes and complications occurrence will be compared.

DETAILED DESCRIPTION:
After a complete ophthalmic evaluation the recruited patients with inactive graves orbitopathy and upper eyelid retraction eligible for the study will be randomly separated in two groups.

The evaluation also includes a face photography in primary position of gaze, a OSDI questionnaire, a quality of life questionnaire, schirmmer test, lissamine green evaluation and eyelid position measurements.

In the first group the patients will be submitted to blepharotomy for surgical correction of their upper eyelid retraction.

In the second group the patients will be submitted to a posterior mullerectomy and gradual recession of the elevator muscle aponeurosis for surgical correction of their upper eyelid retraction.

The outcomes will be compared between the two groups after a 6 month followup.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years old
* controlled thyroid function
* absence of strabismus
* absence of other ocular pathology, such as high myopia
* understanding the protocol and according the terms

Exclusion Criteria:

* pregnancy
* history of previous upper lid surgery
* myasthenia gravis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
clinical measure of the Margin Reflex distance | 6 months
  Assessment of the surgical correction effectiveness by measuring the eyelid lengthening

SECONDARY OUTCOMES:
evaluation of ocular surface with OSDI (Ocular Surface Disease Index) questionnaire, clinical measures with Schirmmer test green lissamine and tear film breakup Time. | 6 months
  OSDI (Ocular Surface Disease Index) is a questionnaire of dry eye symptoms Schirmmer test - measures tear production green lissamine test - evaluate ocular surface damage Tear film Break Up Time - evaluate tear's quality
From the patients digital photographs,computed assisted measurements of eyelid shape and contour will be performed. | 6 months
  with a specific software (contour) the contour and shape of the operated eyelids will be measured.
  Comparison will be made with previous photographs and of normal subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Allan p Goncalves, Dr, Principal Investigator — Staff
Locations (1):
- Hospital das Clinicas - FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Pereira TS, Kuniyoshi CH, Leite CA, Gebrim EMMS, Monteiro MLR, Pieroni Goncalves AC. A Comparative Study of Clinical vs. Digital Exophthalmometry Measurement Methods. J Ophthalmol. 2020 Mar 23;2020:1397410. doi: 10.1155/2020/1397410. eCollection 2020. PMID 32280513
- [Derived] Goncalves ACP, Nogueira T, Goncalves ACA, Silva LD, Matayoshi S, Monteiro MLR. A Comparative Study of Full-Thickness Blepharotomy Versus Transconjunctival Eyelid Lengthening in the Correction of Upper Eyelid Retraction in Graves' Orbitopathy. Aesthetic Plast Surg. 2018 Feb;42(1):215-223. doi: 10.1007/s00266-017-0978-9. Epub 2017 Oct 12. PMID 29026936